CLINICAL TRIAL: NCT01821937
Title: Pharmacokinetics of Single and Multiple Oral Doses of 120 mg and 240 mg BI 201335 in Healthy Chinese Volunteers
Brief Title: Pharmacokinetics of Faldaprevir of Soft Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1220.52
Record Dates: First submitted 2013-03-25; First posted 2013-04-01 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — faldaprevir

ARMS (2):
- faldaprevir(high dose) (Experimental): 10 subjects (approximate sex ration: 1:1) will be assigned to trial by single and multiple dose.
  Interventions: Drug: faldaprevir(high dose)
- Faldaprevir(low dose) (Experimental): 10 subjects (approximate sex ration: 1:1) will be assigned to trial by single and multiple dose.
  Interventions: Drug: Faldaprevir(low dose)

INTERVENTIONS:
Drug: faldaprevir(high dose) — faldaprevir(high dose) will be taken by 1 day single use and 10 days multiple use. the subjects will be assigned to high dose treatment in random order
  Arms: faldaprevir(high dose)
Drug: Faldaprevir(low dose) — faldaprevir(low dose) will be taken by 1 day single use and 10 days multiple use. the subjects will be assigned to low dose treatment in random order
  Arms: Faldaprevir(low dose)

SUMMARY:
The aim of the trial is to assess the bioavailability of Faldaprevir soft capsule with single oral dose and multiple oral doses in Chinese subjects

ELIGIBILITY:
Inclusion criteria:

Healthy male and female subjects

Exclusion criteria:

Any relevant deviation from healthy conditionsAny relevant deviation from healthy conditions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.52.86001 Boehringer Ingelheim Investigational Site, Beijing, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Faldaprevir 120 mg: Oral administration of Faldaprevir 120 mg (BI 201335) soft gel capsule.
  The study was divided into two phases, the first being a single dose and the second a multiple dose.
  During the single dose treatment (days 1-5), subjects received one single dose in the morning of day 1.
  During the multiple dose treatment (days 6-15), subjects received multiple oral doses of faldaprevir once daily from day 6 to day 15.
- Faldaprevir 240 mg: Oral administration of Faldaprevir 240 mg (BI 201335) soft gel capsule.
  The study was divided into two phases, the first being a single dose and the second a multiple dose.
  During the single dose treatment (days 1-5), subjects received one single dose in the morning of day 1.
  During the multiple dose treatment (days 6-15), subjects received multiple oral doses of faldaprevir once daily from day 6 to day 15.
Period: Overall Study
Arm/Group | Faldaprevir 120 mg | Faldaprevir 240 mg
Started | 10 | 15
Completed | 10 | 12 (2 patients discontinued during Single dose period,1 Patient discontinued during Multiple dose period)
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 3

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This set included all 25 subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Faldaprevir 240 mg: Oral administration of Faldaprevir 240 mg (BI 201335) soft gel capsule
  The study was divided into two phases, the first being a single dose and the second a multiple dose.
  During the single dose treatment (days 1-5), subjects received one single dose in the morning of day 1.
  During the multiple dose treatment (days 6-15), subjects received multiple oral doses of faldaprevir once daily from day 6 to day 15.
- Total: Total of all reporting groups
Arm/Group | Faldaprevir 120 mg | Faldaprevir 240 mg | Total
Number analyzed (Participants) | 10 | 15 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.5) | 24.8 (5.7) | 25.0 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax,ss (After Multiple Dosing)
Description: C(max,ss) is defined as maximum measured concentration of Faldaprevir in plasma at steady state over a uniform dosing interval tau.
Time Frame: Before drug administration and 24 hours(h), 48,72,96,120,144,168,192,216,216.5,217,218,219,220,222,224,228, 240 h after first administration of Faldaprevir
Population: Pharmacokinetic analysis set (PKS): This set included all subjects in TS who provided at least one Pharmacokinetic (PK) endpoint and had no important protocol violations relevant to the evaluation of PK and provided no emesis with onset at or before twice the median t max .
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Faldaprevir 120 mg | Faldaprevir 240 mg
Number analyzed (Participants) | 10 | 11
ng/mL | 3270 (44.0) | 14200 (35.5)

2. Primary Outcome: AUC(Tau,ss) (After Multiple Dosing)
Description: AUC(tau,ss) is defined as area under the concentration-time curve of Faldaprevir in plasma at steady state over a uniform dosing interval tau.
Time Frame: Before drug administration and 24 hours(h), 48,72,96,120,144,168,192,216,216.5,217,218,219,220,222,224,228,240 h after first administration of Faldaprevir
Population: Pharmacokinetic analysis set (PKS): This set included all subjects in TS who provided at least one PK endpoint and had no important protocol violations relevant to the evaluation of PK and provided no emesis with onset at or before twice the median t max .
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Faldaprevir 120 mg | Faldaprevir 240 mg
Number analyzed (Participants) | 10 | 11
ng*h/mL | 36200 (48.5) | 199000 (49.5)

3. Secondary Outcome: Cmax (After Single Dosing)
Description: Cmax is defined as maximum measured concentration of Faldaprevir in plasma.
Time Frame: Before drug administration and 0.5 hours(h), 1,1.5,2,3,4,6,8,12,24,48,72,96h after administration of Faldaprevir
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Faldaprevir 120 mg | Faldaprevir 240 mg
Number analyzed (Participants) | 10 | 13
ng/mL | 664 (48.7) | 2060 (44.3)

4. Secondary Outcome: AUC(0-tz) (After Single Dosing)
Description: AUC (0-tz) is defined as area under the concentration-time curve of the analyte in plasma over the respective time interval, where t and z define beginning and end times of the time interval.
Time Frame: Before drug administration and 0.5 hours(h), 1,1.5,2,3,4,6,8,12,24,48,72,96h after administration of Faldaprevir
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Faldaprevir 120 mg | Faldaprevir 240 mg
Number analyzed (Participants) | 10 | 13
ng*h/mL | 14600 (38.9) | 37900 (45.5)

5. Secondary Outcome: t(1/2,ss) (After Multiple Dosing)
Description: t(1/2,ss) is defined as the terminal half-life of Faldaprevir in plasma at steady state.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Faldaprevir 120 mg | Faldaprevir 240 mg
Number analyzed (Participants) | 10 | 11
hour | 31.2 (9.27) | 20.0 (23.6)

6. Secondary Outcome: Tmax,ss (After Multiple Dosing)
Description: tmax,ss is defined as the time from last dosing to the maximum measured concentration of Faldaprevir in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Faldaprevir 120 mg | Faldaprevir 240 mg
Number analyzed (Participants) | 10 | 11
hour | 2.85 (33.6) | 2.44 (29.8)

ADVERSE EVENTS:
Time Frame: From first intake of the trial medication until the end of the trial (Up to Day 16)
Groups:
- Faldaprevir 120 mg Single Dose: Oral administration of Faldaprevir 120 mg (BI 201335) soft gel capsule.
  The study was divided into two phases, the first being a single dose and the second a multiple dose.
  During the single dose treatment (days 1-5), subjects received one single dose in the morning of day 1.
- Faldaprevir 120 mg Multiple Dose: Oral administration of Faldaprevir 120 mg (BI 201335) soft gel capsule.
  The study was divided into two phases, the first being a single dose and the second a multiple dose.
  During the multiple dose treatment (days 6-15), subjects received multiple oral doses of faldaprevir once daily from day 6 to day 15.
- Faldaprevir 240 mg Single Dose: Oral administration of Faldaprevir 240 mg (BI 201335) soft gel capsule
  The study was divided into two phases, the first being a single dose and the second a multiple dose.
  During the single dose treatment (days 1-5), subjects received one single dose in the morning of day 1.
- Faldaprevir 240 mg Multiple Dose: Oral administration of Faldaprevir 240 mg (BI 201335) soft gel capsule
  The study was divided into two phases, the first being a single dose and the second a multiple dose.
  During the multiple dose treatment (days 6-15), subjects received multiple oral doses of faldaprevir once daily from day 6 to day 15.
Arm/Group | Faldaprevir 120 mg Single Dose | Faldaprevir 120 mg Multiple Dose | Faldaprevir 240 mg Single Dose | Faldaprevir 240 mg Multiple Dose
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 7/10 | 10/10 | 13/15 | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120 mg Single Dose (N=10) | Faldaprevir 120 mg Multiple Dose (N=10) | Faldaprevir 240 mg Single Dose (N=15) | Faldaprevir 240 mg Multiple Dose (N=13)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 5 | 8
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 3
Alanine aminotransferase abnormal (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Bile output abnormal (Investigations) | 0 | 1 | 0 | 1
Bile output increased (Investigations) | 0 | 0 | 0 | 1
Bilirubin conjugated abnormal (Investigations) | 0 | 5 | 0 | 6
Bilirubin conjugated increased (Investigations) | 0 | 3 | 1 | 8
Blood bilirubin abnormal (Investigations) | 0 | 6 | 0 | 7
Blood bilirubin increased (Investigations) | 0 | 3 | 1 | 7
Blood bilirubin unconjugated increased (Investigations) | 0 | 8 | 1 | 12
Blood cholesterol abnormal (Investigations) | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase abnormal (Investigations) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase abnormal (Investigations) | 1 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 2
Blood potassium abnormal (Investigations) | 0 | 1 | 0 | 0
Blood triglycerides abnormal (Investigations) | 0 | 0 | 2 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Haptoglobin abnormal (Investigations) | 1 | 0 | 0 | 0
Haptoglobin decreased (Investigations) | 0 | 0 | 1 | 1
Lipase abnormal (Investigations) | 1 | 0 | 1 | 0
Lipase increased (Investigations) | 2 | 1 | 0 | 1
Protein total abnormal (Investigations) | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 1
Total bile acids increased (Investigations) | 1 | 1 | 1 | 2
Urine bilirubin increased (Investigations) | 0 | 0 | 0 | 3
Urobilinogen urine increased (Investigations) | 0 | 0 | 0 | 3
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 3 | 0 | 2
Chromaturia (Renal and urinary disorders) | 0 | 2 | 1 | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Hypomenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.